CLINICAL TRIAL: NCT06586060
Title: Lung Ultrasound Guided Fluid Balance Strategy in Patients with Lung Contusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ibraheem Abdelmageed, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Master Emergency 1
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung Contusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LUS group (Experimental): lung ultrasound guided fluid management guided by B-line score (BLS). In patients with no or mild extravascular lung water (EVLW) increase (BLS = 0-14), a zero fluid balance (FB) will be targeted if no signs of shock are present. In patients with a moderate or severe increase in EVLW (BLS ≥ 15), a daily negative FB of -250 to -1000 mL will be targeted until BLS drops under 15.
  To reach daily targeted FB, furosemide-induced diuresis and RRT will be used. Furosemide will be administrated in a stepwise manner considering the previous furosemide dose and the FB achieved. If the targeted FB is achieved from the first day of diuretic administration, the furosemide dose will be maintained. If FB is outside the targeted range, the furosemide dose will be progressively reduced or increased until the goal is achieved. RRT will be used in patients with moderate and severe EVLW increase (BLS ≥ 15) if the targeted FB cannot be reached despite using the maximum furosemide dose of 800 mg/day.
  Interventions: Other: lung ultrasound guided fluid balance strategy
- control group (Active Comparator): fluid management will be guided to maintain an adequate intravascular volume while minimising weight gain.fluid and diuretics administration will be given according to the clinical judgement of the treating ICU physician. Various parameters will be used to attain this goal based on case-by-case clinical judgment: lung sounds, heart rate, blood pressure, temperature, urine output, FB, lactate, haemoglobin, haematocrit, serum urea, creatinine, sodium, potassium, chloride, and bicarbonate values
  Interventions: Other: usual care guided fluid balance strategy

INTERVENTIONS:
Other: lung ultrasound guided fluid balance strategy — Lung ultrasound (LUS) guided fluid management based on B-Line score assessment using LUS within 24 hours of icu admission and daily thereafter until icu discharge or for up to 14 days after randomization which ever comes first
  In patients with BLS = 0-14, a zero fluid balance (FB) will be targeted if no signs of shock are present. In patients with BLS ≥ 15, a daily negative FB of -250 to -1000 mL will be targeted until BLS drops under 15. To reach daily targeted FB, furosemide-induced diuresis and RRT will be used In case of shocked patients with BLS < 15: they will receive fluid boluses and packed RBCs to achieve a Hb of 10 and a MAP of >65 mmHg.
  In case of shocked patients with BLS ≥ 15: they will start norepinephrine infusion to reach a MAP of >65 mmHg.
  Arms: LUS group
Other: usual care guided fluid balance strategy — fluid balance management will be guided to maintain an adequate intravascular volume while minimising weight gain within 24 hours of icu admission and daily thereafter until icu discharge or for up to 14 days after randomization which ever comes first. Various parameters will be used to attain this goal based on case-by-case clinical judgment: lung sounds, heart rate, blood pressure, temperature, urine output, lactate, haemoglobin, haematocrit, serum urea, creatinine, sodium, potassium, chloride, and bicarbonate values To reach daily targeted fluid balance, furosemide-induced diuresis and RRT will be used
  Arms: control group

SUMMARY:
Lung contusion is caused by blunt chest trauma, explosion injuries or a shock wave associated with penetrating trauma. These injuries damage alveolar capillaries, so blood and other fluids accumulate in the lung tissue. The excess fluid interferes with gas exchange leading to hypoxia To find out whether lung ultrasound as a non-invasive tool can be used to tailor the better fluid balance strategy to achieve higher oxygenation compared to other conventional methods in patients with lung contusion.

The study will evaluate a fluid management protocol for adult patients, based on the daily assessment of B-line score (BLS) using lung ultrasound, compared to usual care. A pre-specified BLS cut-off value of 15 will be used in this study to correct fluid overload After enrolment, patients were randomly assigned to BLS-guided fluid management (active group) or standard care (control group) in a 1:1 ratio, using a computerised random-number generator.

lung ultrasound guided fluid management based on BLS assessment will be conducted within 24 hours of icu admission and daily thereafter until icu discharge or for up to 14 days after randomization which ever comes first In the active group, with every LU examination, patients will be stratified into four classes: no EVLW increase (BLS = 0-4), mild increase (BLS = 5-14), moderate increase (BLS = 15-29), or severe EVLW increase (BLS ≥ 30).

In patients with no or mild EVLW increase (BLS = 0-14), a zero fluid balance (FB) will be targeted if no signs of shock are present. In patients with a moderate or severe increase in EVLW (BLS ≥ 15), a daily negative FB of -250 to -1000 mL will be targeted until BLS drops under 15. To reach daily targeted FB, furosemide-induced diuresis and RRT will be used. Furosemide will be administrated in a stepwise manner considering the previous furosemide dose and the FB achieved. If the targeted FB is achieved from the first day of diuretic administration, the furosemide dose will be maintained. If FB is outside the targeted range, the furosemide dose will be progressively reduced or increased until the goal is achieved. RRT will be used in patients with moderate and severe EVLW increase (BLS ≥ 15) if the targeted FB cannot be reached despite using the maximum furosemide dose of 800 mg/day.

In case of shocked patients with BLS < 15: they will receive fluid boluses and packed RBCs to achieve a Hb of 10 and a MAP of >65 mmHg.

In case of shocked patients with BLS ≥ 15: they will start norepinephrine infusion to reach a MAP of >65 mmHg.

In the control group, fluid management will be guided to maintain an adequate intravascular volume while minimising weight gain. Various parameters will be used to attain this goal based on case-by-case clinical judgment: lung sounds, heart rate, blood pressure, temperature, urine output, FB, lactate, haemoglobin, haematocrit, serum urea, creatinine, sodium, potassium, chloride, and bicarbonate values

Research outcome measures:

1. Primary (main):

   Difference in p-f ratio between the two groups to find out the best strategy for fluid balance for best p-f ratio.
2. Secondary (subsidiary):

Duration of ventilation Duration of ICU stay Duration of hospital stay

DETAILED DESCRIPTION:
Lung contusion is caused by blunt chest trauma, explosion injuries or a shock wave associated with penetrating trauma. These injuries damage alveolar capillaries, so blood and other fluids accumulate in the lung tissue. The excess fluid interferes with gas exchange leading to hypoxia. The pathophysiology of lung contusion includes ventilation / perfusion mismatching, increased intrapulmonary shunting, increased lung water, segmental lung damage, and a loss of compliance.

Fluid replacement is required to ensure adequate blood volume, but this should be done carefully as fluid overload can worsen pulmonary edema, which may be damaging. There may be wheezing, coughing, bronchorrhea and blood-streaked sputum in up to half of cases. There may be hypotension and reduced cardiac output.

Pulmonary contusion results in bleeding and fluid leakage into lung tissue, which becomes rigid and loses its normal elasticity. The water content of the lung increases over the first 72 hours after injury, and may lead to frank pulmonary edema in more serious cases.

Recently lung ultrasound has emerged as golden tool asses over hydration through the B -LINES score Lung ultrasound has the advantages of being safe, non-invasive and already part of different diagnostic algorithm of life threatening conditions with real time detection of increased extravascular lung water and providing a valuable safety threshold to conduct fluid therapy and optimize volume status.

Aim of the study:

To find out whether lung ultrasound as a non-invasive tool can be used to tailor the better fluid balance strategy to achieve higher oxygenation compared to other conventional methods in patients with lung contusion.

The study will evaluate a fluid management protocol for adult patients, based on the daily assessment of B-line score (BLS) using lung ultrasound, compared to usual care. A pre-specified BLS cut-off value of 15 will be used in this study to correct fluid overload.

Type of the study: prospective randomized controlled trial Study Setting: Emergency department at Assiut University Hospital

Study subjects:

1. Inclusion criteria:

   1. poly trauma patients with lung contusion
   2. isolated lung contusion
   3. blunt chest trauma associated with lung contusion
2. Exclusion criteria:

   1. patient refusal
   2. pregnancy
   3. age less than 18.
   4. Patients with known pulmonary conditions that interfere with interpretation of LUS eg: pulmonary fibrosis ,persistent pleural effusion and pnemonectomy .

After enrolment, patients were randomly assigned to BLS-guided fluid management (active group) or standard care (control group) in a 1:1 ratio, using a computerised random-number generator.

3-lung ultrasound guided fluid management based on BLS assessment within 24 hours of icu admission and daily thereafter until icu discharge or for up to 14 days after randomization which ever comes first All patients will be clinically examined daily in the morning and LUS will be performed at bedside with the patient in supine position . the lung will be scanned from the second to fourth intercostal space on the left and from the second to fifth intercostal space on the right at para sternal , mid clavicular , anterior axillary and mid axillary lines .

The focus of the image will be set at the pleural line level and the depth of penetration will be set to 10 cm. The ultrasound equipment will be the GE LOGIQ ® ultrasound system with the curved probe.

B-lines are hyperechoic,comet-tail artefacts, which emerge from the level of the pleural line and move synchronously with lung sliding.

B-lines will be recorded in each intercostal space (28 site of examination ) .the sum of all B lines will produce a score BLS reflecting the extent of extra vascular lung water accumulation Fluid Management In the active group, with every LU examination, patients will be stratified into four classes: no EVLW increase (BLS = 0-4), mild increase (BLS = 5-14), moderate increase (BLS = 15-29), or severe EVLW increase (BLS ≥ 30).

In patients with no or mild EVLW increase (BLS = 0-14), a zero fluid balance (FB) will be targeted if no signs of shock are present. In patients with a moderate or severe increase in EVLW (BLS ≥ 15), a daily negative FB of -250 to -1000 mL will be targeted until BLS drops under 15. To reach daily targeted FB, furosemide-induced diuresis and RRT will be used. Furosemide will be administrated in a stepwise manner considering the previous furosemide dose and the FB achieved. If the targeted FB is achieved from the first day of diuretic administration, the furosemide dose will be maintained. If FB is outside the targeted range, the furosemide dose will be progressively reduced or increased until the goal is achieved. RRT will be used in patients with moderate and severe EVLW increase (BLS ≥ 15) if the targeted FB cannot be reached despite using the maximum furosemide dose of 800 mg/day.

In case of shocked patients with BLS < 15: they will receive fluid boluses and packed RBCs to achieve a Hb of 10 and a MAP of >65 mmHg.

In case of shocked patients with BLS ≥ 15: they will start norepinephrine infusion to reach a MAP of >65 mmHg.

In the control group, fluid management will be guided to maintain an adequate intravascular volume while minimising weight gain. Various parameters will be used to attain this goal based on case-by-case clinical judgment: lung sounds, heart rate, blood pressure, temperature, urine output, FB, lactate, haemoglobin, haematocrit, serum urea, creatinine, sodium, potassium, chloride, and bicarbonate values. Additionally, central venous oxygen saturation, pulse pressure variation and stroke volume variation will be used to assess fluid responsiveness in patients with shock.

Arterial blood gases for p-f ratio will be calculated daily for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. poly trauma patients with lung contusion
2. isolated lung contusion
3. blunt chest trauma associated with lung contusion

Exclusion Criteria:

1. patient refusal
2. pregnancy
3. age less than 18.
4. Patients with known pulmonary conditions that interfere with interpretation of LUS eg: pulmonary fibrosis ,persistent pleural effusion and pnemonectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | once daily at 10 a.m. for 14 days after randomization
  obtained from arterial blood gases

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No